CLINICAL TRIAL: NCT04348617
Title: A Pilot Study " Effect of Acute Exercise on Food Intake and Energy Expenditure Following a Gastric Bypass: A Better Understanding of Weight Maintenance for Better Intervention"
Brief Title: Effect of Acute Exercise on Food Intake and Energy Expenditure Following a Gastric Bypass
Acronym: ExoABari
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universite du Quebec en Outaouais (Other)
Collaborators: University of Ottawa (Other); Université de Sherbrooke (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Aurelie Baillot, Professor, Universite du Quebec en Outaouais
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-31-2020-323
Record Dates: First submitted 2020-03-26; First posted 2020-04-16 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Appetite; Food intake; Energy expenditure; Food reward; Appetite hormones; Inflammatory response; acute exercise
MeSH Terms: conditions — Obesity | interventions — Walking; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Participants will take part in a randomized exercise and control (rest) condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-Rest (Experimental): This group will perform the exercise condition at least 1 week after the preliminary visit and will perform the resting condition a minimum of 15 days and a maximum of 2 months after the exercise condition.
  Interventions: Other: Moderate exercise; Other: Rest
- Rest-Exercise (Experimental): This group will perform the resting condition at least 1 week after the preliminary visit and will perform the exercise condition a minimum of 15 days and a maximum of 2 months after the resting condition.
  Interventions: Other: Moderate exercise; Other: Rest

INTERVENTIONS:
Other: Moderate exercise — 50 minutes of moderate exercise on treadmill
  Other Names: Walking
Other: Rest — 50 minutes of rest or sedentary activity

SUMMARY:
This pilot study will use a crossover design to explore the effects of acute exercise following bariatric surgery on food intake, energy expenditure, appetite, food reward, appetite hormones, and inflammatory response. Participants will take part in a moderate-intensity exercise session and control condition of 50 minutes. The energy balance will be assessed for 3 days following the condition by giving the participants all the food they can consume for 3 days and having them wear an accelerometer.

The investigators hypothesize that post-gastric bypass participants with higher weight regain will have a higher compensation in response to exercise, thus an increase in food intake and/or a decrease in total energy expenditure after exercise compared to participants with less weight regain; also post-gastric bypass participants with a higher weight regain will have a lower inflammatory response to exercise compared to the group with less weight regain.

DETAILED DESCRIPTION:
Objectives.

1. Explore the feasibility of a multicenter study in post-GB patients;
2. Explore the effects of acute exercise on food intake and energy expenditure post-GB;
3. Explore the effects of acute exercise on the hormonal and inflammatory response post-exercise.

This pilot study will employ crossover design. The Behavioural and Metabolic Research Unit (BMRU) at the School of Human Kinetics of the University of Ottawa will coordinate and standardize the project between the sites. The participants will need to go 5 times to one of the 3 evaluation sites (University of Ottawa: BMRU, Montreal: University of Montreal, School of kinesiology and physical activity or University of Sherbrooke: Research Aging Center of CIUSSS - CHUS).

Considering this is a pilot project, no sample size calculations were conducted. Based on existing studies, 30 participants should be sufficient to achieve the preliminary objectives of this study.

The participants will be asked to present themselves at the evaluation centre on 5 occasions (1 preliminary, 2 experimental, 2 to return leftovers and accelerometers).

During the visits 1, 2 and 4 (1 preliminary and 2 experimental (exercise and control)), the participants will arrive at 7:00 a.m. at the laboratory after 12 hours nocturnal fast. At 9:00 a.m., they will consume a standardized personalized breakfast. Participants will choose themselves the breakfast they want from a validated menu. They will be informed that they can consume the desired quantity of each product; the quantities will be measured to assure the breakfast for the other visits is identical.

During the 1st session, depressive symptoms, the body composition (DEXA), resting metabolic rate and anthropometrics (weight, height, waist circumference) will be measured before breakfast. Afterwards, their socio-demographic information, motivation to eat and binge eating behaviors will be assessed. At 10:30 a.m., participants will perform submaximal exercise for 30 minutes to familiarize themselves with the treadmill, determine the speed and incline of the treadmill to achieve 55% estimated HRR and obtain an estimation of EE during the experimental condition. Subsequently to the first visit, the participants will wear an accelerometer for 7 days and bring it back for the 2nd visit. The day before the 2nd visit, the participants will fill out a food intake journal of the last 24 hours in order to consume the exact same foods (items, quantities and timeframe) the day before the 3rd session.

At least one week after the 1st session, participants will present themselves to the evaluation site for the 2nd session to take part in one of the 2 experimental conditions (control and exercise), which will be randomly assigned and spaced a minimum of 15 days and a maximum of 2 months, yet to be performed the same day of the week. Women will only be tested between day 1 and 8 of their follicular phase. During the experimental conditions, participants will perform exercise on a treadmill (50 minutes at 55% of estimated HRR) (exercise condition) or the controlled condition (inactive period of calm and stress-free reading) at 10:30 a.m. Sixty minutes following exercise or the inactive period, an ad libitum buffet will be served to assess caloric and macro-nutritional intake. Appetite sensations will be assessed in the morning during fasting, before/after exercise, before/after ad libitum buffet as well as 1 and 2 hours after eating. Food rewards will be measured before and 1 hour after the meal. Blood samples will be collected 5 times by a nurse after a catheter has been installed, representing a total of 108 ml of blood collected (morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before the buffet) to analyze appetite-related hormones (ghrelin, peptide YY (PYY) and glucagon-like peptide-1 (GLP-1)) and inflammatory parameters (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1). Finally, participants will wear an accelerometer (Actigraph® GT3X+) for 3 days following the sessions to determine their total EE outside of the laboratory. They will also leave with 3 days' worth of meals of their choice and will need to bring back any leftovers in order to calculate their caloric intake.

In the exercise condition, a 50-minute effort at 55% of the estimated HRR will be performed on the treadmill following a 3-minute warm-up at 2.5 km/h and will be followed by a 2-minute active recovery period at 2.5 km/h then sitting for 3 minutes. The estimated maximum heart rate will be calculated from the most accurate prediction equation for a population with obesity: 208 - 0.7 × age. The heart rate will be monitored with a heart rate monitor throughout the exercise and recovery to ensure that the intensity of the exercise is maintained.

The energy intake and macronutrients from the ad libitum will be measured with the validated technique of the food menu. A total of 62 items will be on the menu to ensure that sufficient hot meals, snacks, fruits, vegetables and beverages are available to the participants. Briefly, participants will be invited to choose from this validated menu, their breakfast, the meals they would like to have for lunch and after lunch the meals they would like to eat for the next 3 days (from midnight to midnight). The research assistant/student will instruct them to consume as much of these products as they want. All selected foods will be prepared and measured according to the guidelines described above (34). The food and beverages selected for the 3 days will be packed in plastic containers or bottles, which will be placed in a portable cooler for the participants to take with them. They must return all leftovers in their original containers. The selected and prepared foods will be weighted to the nearest gram using an electronic food scale before being consumed or placed in coolers. The macronutrient composition of foods and beverages consumed will be determined and analyzed in Ottawa using Food Processor SQL software (version 9.6.2; ESHA Research).

Appetite and satiety will be measured using a computer-based visual analogue scale (VAS) (0-100mm). The desire to eat, hunger, satiety and potential food consumption will be assessed. The level of satiety will be evaluated using the "satiety quotient" method adapted from Green et al, which quantify variations in subjective appetite measurements (mm) for each 100kcal of food consumed. The Leeds Food Preference Questionnaire (LFPQ) will be used to assess food reward, i.e. explicit food pleasure and implicit and explicit food motivation.

Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The blood plasma samples collected for hormone analysis (ghrelin, PYY, GLP-1) will be collected in EDTA tubes. Immediately after blood sampling, a precise protocol will be used for each targeted hormone to preserve their integrity.

ELIGIBILITY:
Inclusion Criteria:

* declare to be an adult (≥ 18 years old)
* self-declared physically inactive (practicing less than 150 min/week of moderate to high intensity physical activity)
* received a gastric bypass Roux-en-Y more than 24 months ago at the Ottawa Hospital
* have regained weight ≤5%/year of total weight loss at nadir or ≥15%/year (n=15 regain)

Exclusion Criteria:

* be pregnant, breastfeeding or menopausal
* have depressive symptoms (score ≥16 at the Center Epidemiologic Depression-Scale)
* take medication that may influence appetite or weight loss
* declare they cannot walk for 50 minutes
* be classified as high risk according to the stratification model of the ACSM (people with heart disease, Peripheral vascular or cerebrovascular disease, chronic obstructive pulmonary disease, asthma, interstitial lung disease or cystic fibrosis, type 1 and 2 diabetes, thyroid disorders, kidney or liver disease) and not having medical authorization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of energy intake between rest and exercise conditions (kcal/d) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  The energy intake and macronutrients from the ad libitum will be measured with the validated technique of the food menu. A total of 62 items will be on the menu to ensure that sufficient hot meals, snacks, fruits, vegetables and beverages are available to the participants. Briefly, participants will be invited to choose from this validated menu, their breakfast, the meals they would like to have for lunch and after lunch the meals they would like to eat for the next 3 days (from midnight to midnight). The research assistant will instruct them to consume as much of these products as they want. All selected foods will be prepared and measured according to the guidelines described above. The food and beverages selected for the 3 days will be packed in plastic containers or bottles, which will be placed in a portable cooler for the participants to take with them. They must return all leftovers, packaging and peels in their original containers.
Change of total energy expenditure post-experimentation between rest and exercise conditions (kcal/d) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Total energy expenditure: Using an accelerometer (Actigraph® GT3X+) worn on the right side at the waist for 3 days following the experimental conditions (except during showering and aquatic physical activities), total EE will be estimate (ActiLife® Software). In parallel, the participant will have to complete a physical activity logbook during the 3 days of wearing the accelerometer.

SECONDARY OUTCOMES:
Change of appetite sensation score during experimentation and between conditions; visual analog scale (0-100mm) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Appetite and satiety will be measured using a computer-based visual analogue scale (VAS) (0-100mm) in the morning during fasting, before/after exercise, before/after ad libitum buffet as well as 1 and 2 hours after eating. The desire to eat, hunger, satiety and potential food consumption will be assessed using the following questions: 1) "How intense is your desire to eat?" (Very weak - very strong); 2) "How hungry are you?" Not at all hungry - as hungry as ever); 3) "How full are you feeling?" (Not at all - Completely), and 4) "How much food do you think you can eat?" (Nothing at all - A large quantity). Higher scores mean higher desire to eat, appettite, and a lower satiety.
Change of food rewards score during experimentation and between conditions, The Leeds Food Preference Questionnaire | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  The Leeds Food Preference Questionnaire (LFPQ) will be used before and 1 hour after the meal during the experimental conditions to assess food reward, i.e. explicit food pleasure and implicit and explicit food motivation. This questionnaire is a validated computerized procedure, during which 16 personalized different food images will be presented to participants for approximately 10 minutes. Food images were previously classified according to fat content (rich vs. low) and/or taste (salty vs. sweet) to form four categories: high fat and salt, low fat and salt, high fat and sugar, and low fat and sugar.
Change of blood IL-6 concentration during experimentation and between conditions | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Baseline resting energy expenditure (kcal/d) | Baseline
  Resting energy expenditure will be evaluated by indirect calorimetry with continuous evaluation of O2 and CO2 sampled with a transparent hood, after calibration of the gas analyzers.
Exercise energy expenditure (kcal/d) | Baseline and during the exercise condition = at least one week after baseline evaluation (visit 2) OR 15 days to a maximum of 2 months after visit 2
  Exercise energy expenditure will be evaluated by indirect calorimetry with continuous evaluation of O2 and CO2 sampled with a mouthpiece, after calibration of the gas analyzers.
Change of blood ghrelin concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The blood plasma samples collected for ghrelin analysis will be collected in EDTA tubes. Immediately after blood sampling, a precise protocol will be used to preserve their integrity. The analysis of ghrelin will be carried out with ELISA kits specific to ghrelin: Millipore, Etobicoke, ON, Canada. Blood samples will be collected 5 times during the experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood Glucagon-like peptide-1 (GLP-1) concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The blood plasma samples collected for GLP-1 analysis will be collected in EDTA tubes. Immediately after blood sampling, a precise protocol will be used to preserve their integrity. The analysis of GLP-1 will be carried out with ELISA kits specific to ghrelin: Linco Research, St Louis, MO, USA. Blood samples will be collected 5 times during the experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood peptide YY (PYY) concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The blood plasma samples collected for PYY analysis will be collected in EDTA tubes. Immediately after blood sampling, a precise protocol will be used to preserve their integrity. The analysis of PYY will be carried out with ELISA kits specific to PYY: Linco Research, St Louis, MO, USA. Blood samples will be collected 5 times during the experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Baseline Kg of fat free mass; Dual Energy X-ray Absorptiometry | Baseline
  It will be evaluated by Dual Energy X-ray Absorptiometry.
Baseline Eating behavior score; The Three Factor Eating Questionnaire | Baseline
  The Three Factor Eating Questionnaire, also called Eating Inventory, developed by Stunkard et Messick will be used to identify different eating behaviours or motivations to eat. This 51-question, self-administered questionnaire identifies three "factors": cognitive restraint (21 questions) which measures dietary self-regulation; disinhibition (16 questions) which assesses loss of control over eating and susceptibility to hunger (14 questions), which describes subjective feelings of hunger and cravings.All TFEQ items are coded with either 0 or 1 point leading to maximum sum scores of 21 points for the domain of 'cognitive restraint', 16 points for 'disinhibition' and 14 points for 'hunger'. Higher scores indicate stronger characteristic values in the domains.
Presence of binge eating behaviors; Eating Disorder Examination Questionnaire and Binge Eating Scale | Baseline
  The first section of the Eating Disorder Examination Questionnaire consists of 22 items that allow participants to record the frequency and intensity with which they adopted inappropriate attitudes and behaviours over the past four weeks. A score greater than or equal to 4 is considered clinically significant and suggests a diagnosis of an eating disorder.
  The Binge Eating Scale is a validated 16-item self-administered questionnaire. For each item, the participant must choose from several sentences the wording that best corresponds to their current situation. The score can vary between 0 and 3 or between 0 and 2 for each item. A total score (obtained from the sum of the scores of each of the 16 items) greater than or equal to 18 indicates significant binge eating behaviors.
Baseline Kg of fat mass | Baseline
  It will be evaluated by Dual Energy X-ray Absorptiometry.
Baseline total energy expenditure | Baseline
  Using an accelerometer (Actigraph® GT3X+) worn on the right side at the waist for 7 days after the preliminary visit (except during showering and aquatic physical activities), total EE will be estimate (ActiLife® Software). In parallel, the participant will have to complete a physical activity logbook during the 7 days of wearing the accelerometer.
Change of blood IL-10 concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood IL-1ra concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood IL-8 concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood TNF-α concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood sTNFR concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood MIP-1β concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.
Change of blood MCP-1 concentration during experimentation and between conditions (pg/ml) | At least one week after baseline evaluation (visit 2) and 15 days to a maximum of 2 months after visit 2
  Blood samples taken with a catheter placed in the anterior ulnar vein of the dominant arm will be collected by a qualified nurse. The inflammatory profile (IL-6, IL-10, IL-1ra, IL-8, TNF-α, sTNFR, MIP-1β, MCP-1) will be evaluated with X-Map technology using Luminex 200 (EMD Millipore, Burlington, MA, USA). Blood samples will be collected 5 times during each experimental visits: morning during fasting, before/after exercise or control condition, 30 minutes after exercise or control condition and before lunch.

CONTACTS AND LOCATIONS:
Locations (1):
- Aurelie Baillot, Gatineau, Quebec, Canada